CLINICAL TRIAL: NCT03409068
Title: The Effectiveness of C2-C4 Compartment Block Versus Block of Costagliola, in the Control of Persistent Postoperative Pain in Patients Undergoing Carotid Thromboendarterectomy
Brief Title: C2-C4 Compartment Block Versus Block of Costagliola, in TEAC
Acronym: TEAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Salvatore Hospital of L'Aquila (Other)
Responsible Party: Principal Investigator, Emiliano Petrucci, Medical Doctor, San Salvatore Hospital of L'Aquila
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 0174363/2017
Record Dates: First submitted 2018-01-17; First posted 2018-01-24 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Somatic Pain; Neuropathic Pain
Keywords: Carotid thromboendarterectomy; Carotidodynia
MeSH Terms: conditions — Nociceptive Pain; Neuralgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- C2-C4 compartment block (Experimental): Experimental: the C2-C4 compartment anesthetic block is performed by injecting Levobupivacaine 0.375% 20 mL between the posterior face of the middle scalenous muscle, the anterior face of the posterior scalene muscle and the lower plane of the sternoscleidomastoid muscle.
  Interventions: Procedure: C2-C4 compartment anesthetic block
- Costagliola block (Active Comparator): Active Comparator: the Costagliola anesthetic block is performed by injecting Levobupivacaine 0.375% 20 mL injected in the posterior margin of the sternocleidomastoid muscle and along the anterior border of the same muscle.
  Interventions: Procedure: Costagliola block

INTERVENTIONS:
Procedure: C2-C4 compartment anesthetic block — C2-C4 compartment anesthetic block is performed by injecting levobupivacaine 0.375% 20 mL between the posterior face of the middle scalenus muscle, the anterior face of the posterior scalene muscle and the lower plane of the sternoscleidomastoid muscle.
  Other Names: Intermediate cervical plexus block
  Arms: C2-C4 compartment block
Procedure: Costagliola block — Costagliola block is performed by injected by injecting levobupivacaine 0.375% 20 mL along the anterior and the posterior border of sternocleidomastoid muscle
  Other Names: Superficial cervical plexus block
  Arms: Costagliola block

SUMMARY:
C2-C4 compartment block compared to the Costaiola block, in the control of persistent postoperative pain (somatic and neuropathic) in patients undergoing carotid thromboendarterectomy

DETAILED DESCRIPTION:
A comparative analysis will assess the somatic pain (scores ≥4 on the NRS scale) and neurapathic pain (by the Lindblom roller and Von Frei hair tests) between group A (block group of the C2-C4 compartment ) and the control group B (block group according to Costagliola), during the 3 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing to carotid thromboendarterectomy

Exclusion Criteria:

* ASA status: 4
* pregnancy
* BMI > 39,99
* neurological impairment
* neck anatomical abnormalities
* status of sepsis
* coagulopathy
* neck cancer
* neck infections

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2019-01-18 (Actual)

PRIMARY OUTCOMES:
somatic pain | 3 mounths after surgery
  Somatic pain assessed by Numeric Pain Rating Scale for pain (the 11-point numeric scale ranges from '0' representing "no pain" to '10' representing the "worst pain imaginable"

SECONDARY OUTCOMES:
Opiates request | 3 mounths after surgery
  Request of opiates, assessed in mg of equianalgesic dose of morphine after 3 mouths from surgery
Pregabalin request | 3 months
  Pregabalin request in mg, 3 months after surgery
Neuropathic pain | 3 months
  Presence of neuropathic disturbances, assessed with von Frey hair test and Lindblom test

CONTACTS AND LOCATIONS:
Overall Officials: Emiliano Petrucci, MD, Principal Investigator — SS Filippo and Nicola Academic Hospital of Avezzano
Locations (1):
- SS Filippo and Nicola Academic Hospital of Avezzano, Avezzano, L'Aquila, Italy

IPD SHARING:
Plan to Share IPD: No